CLINICAL TRIAL: NCT05017922
Title: Efficacy of TACE Combined With Endoscopic Therapy for Unresectable Hepatocellular Carcinoma With Esophagogastric Varices
Brief Title: Efficacy of TACE With Endoscopic Therapy for Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021719-Tao
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma; Esophagogastric Varices
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined group (Experimental): unresectable hepatocellular carcinoma patients who received TACE plus endoscopic therapy
  Interventions: Procedure: transarterial chemoembolization combined with endoscopic therapy
- control group (Other): unresectable hepatocellular carcinoma patients who only received TACE
  Interventions: Procedure: transarterial chemoembolization combined with endoscopic therapy

INTERVENTIONS:
Procedure: transarterial chemoembolization combined with endoscopic therapy — TACE: The tip of the catheter was advanced into tumor-feeding artery based on the tumor location and size. 5-Fu was injected. Then the chemolipiodolization was performed, using oxaliplatin, epirubicin and lipiodol. If stagnant flow did not realized, then injected pure lipiodol. If the tumor-feeding artery still cannot be completely embolized, several absorbable gelatin sponge particles would be injected. Endoscopic therapy: After the site of esophageal varices was identified by the gastroscopy, spiral ligation using the EVL device (COOK, MBL-6-F) was performed and ensure the varices were fully inhaled, 1-3 rubber bands were used totally. After EVL, water was sprayed to the ligation sites to check for bleeding. If gastric varices were found, EIS was performed using the 'sandwich method' of hypertonic glucose-tissue adhesive-normal saline. Make sure the needle entered the varieose vein before inject drugs, and repeated the injection if necessary.

SUMMARY:
The study is aimed to explore the efficacy of transarterial chemoembolization (TACE) combined with endoscopic therapy for unresectable hepatocellular carcinoma (HCC) complicated with esophagogastric varices (EGV) and seek out predictors associated with survival.

ELIGIBILITY:
Inclusion Criteria:

* 1. HCC was diagnosed in accordance with the 2017 edition of diagnosis guidelines, all patients were in CNLC stage Ib to IIIa, and treated with TACE; 2. EGV was demonstrated through endoscopic examination; 3. Child-Pugh grade A or B, or grade C patients improved liver function to grade A or B through aggressive treatment; 4. age between 18 and 75 years.

Exclusion Criteria:

* 1. HCC with diffuse or distant metastasis, or with other systemic malignancies; 2. severe jaundice, hepatic encephalopathy, refractory ascites or hepatorenal syndrome; 3. severe cardiac, cerebrovascular, lung and renal diseases and cannot tolerate endoscopic treatment; 4. severe coagulation dysfunction; 5. severe infection, bleeding with unstable vital signs; 6. history of liver surgery; 7. cannot or refuse to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Time of overall survival | In July 2020 or the day of death or the day of lost to follow-up or follow-up for 3 years
  Differences of overall survival between two groups
Number of bleeding episodes | In July 2020 or the day of death or the day of lost to follow-up or follow-up for 3 years
  Differences of bleeding episodes between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital , Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Tao Z, Ruan Y, Peng Z, Zhang K, Gao Y. Transarterial Chemoembolization Combined With Endoscopic Therapy Is Beneficial for Unresectable Hepatocellular Carcinoma With Esophagogastric Varices. Front Oncol. 2021 Dec 2;11:783574. doi: 10.3389/fonc.2021.783574. eCollection 2021. PMID 34926300